CLINICAL TRIAL: NCT07389005
Title: Timed Exercise in Prediabetes With Extreme Chronotype
Brief Title: Exercise, Chronotype, and Prediabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REALIGN
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes; Overweight , Obesity
Keywords: Prediabetes; Overweight; Obesity; Exercise; Chronotype
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will receive a code so that the person in charge with the data quality check and data analyses will be blinded to the interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AM exercise (Experimental): Behavioral: Timing of exercise
  Interventions: Behavioral: Timing of exercise
- PM exercise (Experimental): Behavioral: Timing of exercise
  Interventions: Behavioral: Timing of exercise
- Control (Active Comparator): Behavioral: Control
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Timing of exercise — An acute exercise bout of cycling performed in the morning at 9 AM
  Arms: AM exercise
Behavioral: Timing of exercise — An acute exercise bout of cycling performed in the morning at at 5 PM
  Arms: PM exercise
Behavioral: Control — No exercise
  Arms: Control

SUMMARY:
The goal of this clinical trial is to find out whether exercising at the right time of day, based on a person's natural body clock, leads to greater health benefits in people living with prediabetes. The main question it aims to answer is whether doing a single session of exercise in the morning or in the evening affects how the body handles sugar differently in adults with prediabetes who have an extreme natural body clock. This will be done by comparing three conditions (no-exercise, morning exercise, and evening exercise) within the same participant. Each condition will be tested on a different day, with at least 14 days between the test days. During the no-exercise test days, participants will come to the study centre and will only be allowed to do sedentary activities (e.g. office work, reading, or screen time). During the morning exercise test days, participants will perform an exercise session at 9:00 am that involves short periods of very hard effort followed by short rest periods. Whereas for the evening exercise test days, the same type of exercise will be performed at 5:00 pm.

DETAILED DESCRIPTION:
Chronotype refers to an individual's circadian preferences for being active and fully functional at certain times of the day. Using validated questionnaires, individual's chronotype can be categorized to either a morning (lark), evening (owl), or intermediate (neutral) chronotypes. Individuals with morning chronotype wake up and go to bed early. Therefore, their calorie distribution as well as peak mental and physical performances predominantly occur earlier in the day. This is in contrast with individuals with evening chronotype that wake up and go to bed late, resulting in most of their calorie consumption happens later in the day. They are also more active and alert in the evening. Growing evidence has shown that late afternoon or evening exercise is better than morning exercise for blood glucose control in individuals with type 2 diabetes (T2D) or those at risk of T2D. In men with T2D, two weeks of high-intensity interval training (HIIT) reduced continuous glucose monitor (CGM)-based glucose concentration when performed in the afternoon than in the morning. This finding was further supported by a retrospective study involving men at risk for or T2D that found afternoon exercise led to superior peripheral insulin sensitivity, insulin-mediated suppression of adipose tissue lipolysis, and fasting plasma glucose. Interestingly, in a recently published crossover trial involving men and women, with and without T2D, no difference was observed in 24-hour glucose profile assessed using CGM across all cohorts (including gender and diabetes status) between morning and evening exercise. However, morning exercise increased post-exercise blood glucose levels during the two hours recovery period in both men and women with T2D, which was not observed following the evening exercise. It is important to note that all the above-mentioned studies are either excluding individuals with extreme chronotype or the chronotype of the participants was not clearly reported. This limitation raises an important research question: Do people living with extreme chronotype respond differently to timed exercise? Therefore, in this study, it is hypothesize that people living with prediabetes and extreme chronotype will gain superior metabolic benefits when the timing of exercise is aligned with their chronotype. To test this, a randomized controlled cross-over study is conducted in which participants are subjected to three conditions that are no-exercise, morning exercise, and evening exercise. The main outcome is insulin sensitivity determined by a 2-step hyperinsulinemic-euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated written informed consent prior to any study specific procedures
2. Adult men and women aged between more than 18 and ≤ 75 years
3. Body mass index (BMI) of 25 - 35 kg/m2
4. Stable weight (no weight loss or gain > 3 kg in the past 3 months)
5. Pre-diabetes defined as an isolated impaired glucose tolerance or a combination of impaired glucose tolerance and impaired fasting glucose (values are based on the American Diabetes Association (ADA):

   1. impaired glucose tolerance (plasma glucose 140 mg/dL to 199 mg/dL, 120 minutes after consumption of 75g of glucose)
   2. impaired fasting glucose (fasting plasma glucose 100 mg/dL to 125 mg/dL)
6. Morning (Morningness-Eveningness Questionnaire [MEQ] score ≥ 59) or evening (MEQ score ≤ 41) chronotype

Exclusion Criteria:

1. Previously diagnosed with type 2 diabetes
2. Moderate to severe anemia (hemoglobin < 10 g/L)
3. Uncontrolled hypertension
4. Abnormal electrocardiogram (ECG) at rest judged by the study physician
5. Pregnancy or breastfeeding
6. HIV, hepatitis B, or C infection
7. Disorders of blood clotting or wound healing
8. Positive history of venous thrombosis (contraindication for clamp)
9. Hypersensitivity to local anesthetics (contraindication for fat/muscle biopsies)
10. Night shift work in the last 3 months
11. Travel across > 1 time zone in the last 3 months
12. Participation in another clinical trials that may possibly hamper the study results
13. Engagement in structured exercise activities > 2 hours a week
14. Any acute condition, exacerbation of chronic condition, or medical history that in the investigator's opinion would interfere with the study
15. Any contraindication for MRI scanning
16. Medication use known to hamper safety during the study procedures
17. Non-German speaking

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on insulin sensitivity assessed using insulin sensitivity index (reported as M-value: mg x kg-1 x min-1) during an hyperinsulinemic-euglycemic clamp

SECONDARY OUTCOMES:
Skeletal muscle metabolites | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on skeletal muscle mitochondrial respiration (pmol/mg/s) measured with high resolution respirometry
Skeletal muscle clock genes | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on quantified DNA measured with quantitative polymerase chain reaction (qPCR)
Adipose tissue metabolites | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on adipose tissue mitochondrial respiration (pmol/mg/s) measured with high resolution respirometry
Adipose tissue clock genes | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on quantified DNA measured with quantitative polymerase chain reaction (qPCR)
Hepatic glycogen content assessed using 13C Magnetic Resonance Spectroscopy | Post-dinner on exercise day
  Effect of timed exercise on hepatic glycogen content, expressed in millimoles per liter (mmol/L) of liver tissue
Serum glucose | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on serum glucose levels (mg/dL) determined from venous blood draws
Serum free fatty acids | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on serum free fatty acid levels (mmol/L) determined from venous blood draws
Serum triglycerides | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on serum triglycerides (mg/dL) determined from venous blood draws
Serum cholesterol | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on serum cholesterol (mg/dL) determined from venous blood draws
Serum insulin | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on serum insulin levels (uIU/mL) determined from venous blood draws
Resting energy expenditure assessed using indirect calorimetry | 12 to 24 hours post-exercise intervention
  Effect of timed exercise on resting energy expenditure, expressed in kilocalories per day (kcal/day)
Objective sleep quantity and quality assessed using an actighrapy device | The nighttime of exercise intervention day
  Effect of timed exercise on sleep duration, efficiency, and fragmentation are measured objectively from the actighrapy device

OTHER OUTCOMES:
Liver lipid content measured using ¹H/³¹P Magnetic Resonance Spectroscopy | Baseline assessment
  To assess the difference in liver lipid content in percentage (%) between morning versus evening chronotypes
Skeletal muscle lipid content measured using ¹H/³¹P Magnetic Resonance Spectroscopy | Baseline assessment
  To assess the difference in skeletal muscle lipid content in percentage (%) between morning versus evening chronotypes
Body composition expressed as fat mass (kg and %) and fat-free mass (kg) assessed using Bodpod and Bioelectrical Impedance | Baseline assessment
  To assess the difference in body composition between morning versus evening chronotypes
Maximal aerobic capacity measured using spiroergometry | Baseline assessment
  To assess the difference in maximal aerobic capacity (VO₂max) between morning versus evening chronotypes
Subjective sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI) | Baseline assessment
  To assess the difference in subjective sleep quality between morning versus evening chronotypes. Total score range of 1 to 21, higher scores indicating poorer sleep quality
Level of sleepiness assessed using the Stanford Sleepiness Scale (SSS) | Baseline assessment
  To assess the difference in level of sleepiness between morning versus evening chronotypes. On a 7-point scale, 1 representing feeling alert and 7 indicating being almost in reverie
Consumption of specific foods or food groups assessed using the DEGS1-Food Frequency Questionnaire (FFQ) | Baseline assessment
  To assess the difference in consumption frequency of specific foods or food groups (expressed as times per week) between morning versus evening chronotypes
Hedonic hunger assessed using the Power of Food Scale questionnaire | Baseline assessment
  To assess the difference in hedonic hunger between morning versus evening. Mean score of 15 items rated on a 5-point Likert scale (range 1-5). Higher scores indicate greater psychological responsiveness to food cues
Severity and type of food cravings assessed using the Control of Eating Questionnaire (CoEQ) | Baseline assessment
  To assess the difference in self-reported craving strength between morning versus evening chronotypes. A numeric rating scale ranges from 0 to 10. Higher scores indicate stronger food cravings
Subjective physical activity levels determined using the International Physical Activity Questionnaire (IPAQ) | Baseline assessment
  To assess subjective physical activity levels (low, moderate, high expressed as MET-minutes/week) between morning versus evening chronotypes
Cognitive performance assessed using the Sustained Attention to Response Test (SART) | Baseline assessment
  To assess the difference in cognitive performance between morning versus evening chronotypes. Performance is assessed using commission errors (incorrect responses to no-go stimuli), omission errors (missed responses to go stimuli), mean reaction time, and reaction time variability, with higher error rates and greater reaction time variability indicating poorer sustained attention and inhibitory control
Cognitive performance assessed using the Brief Psychomotor Vigilance Test (PVT-B) | Baseline assessment
  To assess the difference in cognitive performance between morning versus evening chronotypes. Performance is assessed using mean reaction time, number of lapses (reaction times ≥500 ms), and fastest 10% reaction times, with slower reaction times and more lapses indicating reduced vigilant attention and alertness.
Well-being assessed using the World Health Organization-Five Well-being Index (WHO-5) | Baseline assessment
  To assess the difference in well-being between morning versus evening chronotypes. Scores range from 0 to 25 with higher scores indicating better well-being and psychological health
Mental health assessed using the Patient Health Questionnaire-9 (PHQ-9) | Baseline assessment
  To assess the difference in mental health between morning versus evening chronotypes. A 9-item self-report questionnaire assessing depressive symptoms over the past two weeks, scored from 0 to 27 with higher scores indicating greater severity of depressive symptoms
Quality of life assessed using the 36-Item Short Form Survey Instrument (SF-36) | Baseline assessment
  To assess the difference in quality of life between morning versus evening chronotypes. A self-report questionnaire assessing health-related quality of life across eight domains-physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health-with scores transformed to a 0-100 scale, where higher scores indicate better health and functioning

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center (DDZ), Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No
Participant data will only be discussed with other researcher on group level. We are not interested in sharing individual participant data.

REFERENCES:
- [Background] Keller MJ, Brady AJ, Smith JAB, Savikj M, MacGregor K, Jollet M, Oberg SB, Nylen C, Bjornholm M, Rickenlund A, Carlsson M, Caidahl K, Krook A, Pillon NJ, Zierath JR, Wallberg-Henriksson H. Inflammatory markers and blood glucose are higher after morning vs afternoon exercise in type 2 diabetes. Diabetologia. 2025 Sep;68(9):2023-2035. doi: 10.1007/s00125-025-06477-5. Epub 2025 Jun 28. PMID 40580209
- [Background] Mancilla R, Brouwers B, Schrauwen-Hinderling VB, Hesselink MKC, Hoeks J, Schrauwen P. Exercise training elicits superior metabolic effects when performed in the afternoon compared to morning in metabolically compromised humans. Physiol Rep. 2021 Jan;8(24):e14669. doi: 10.14814/phy2.14669. PMID 33356015
- [Background] Savikj M, Gabriel BM, Alm PS, Smith J, Caidahl K, Bjornholm M, Fritz T, Krook A, Zierath JR, Wallberg-Henriksson H. Afternoon exercise is more efficacious than morning exercise at improving blood glucose levels in individuals with type 2 diabetes: a randomised crossover trial. Diabetologia. 2019 Feb;62(2):233-237. doi: 10.1007/s00125-018-4767-z. Epub 2018 Nov 13. PMID 30426166